CLINICAL TRIAL: NCT04279665
Title: Use of Virtual Reality to Reduce Intra-procedural Anxiety and Sedation Needs During Procedures Involving no or Minimal Sedation
Brief Title: Virtual Reality to Reduce Intra-procedural Anxiety and Sedation Needs During Procedures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Equipment changed
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Suraj Kapa, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-005788
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects undergoing electrophysiology procedure (Experimental): Subjects will wear a virtual reality (VR) headset for a total of 40 minutes separated over 2 sessions during an electrophysiology procedure they are already scheduled to undergo.
  Interventions: Device: Virtual Reality (VR)

INTERVENTIONS:
Device: Virtual Reality (VR) — 20 minutes of wearing a virtual reality headset with a choice of 4 environments based on their preference and another 20 minutes with a less immersive condition

SUMMARY:
Researchers are assessing whether use of a virtual reality experience, used during the procedure, can reduce anxiety and improve satisfaction related to the procedure, especially when no or little sedation is being used.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing invasive EP procedures with plan for no or minimal conscious sedation

Exclusion Criteria:

* Patients unable to consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Subject anxiety | 20 minutes
  Measured using a survey question asking participants to rank their anxiety level over the last 20 minutes using a scale of 5 being extremely good (ie, less anxiety); 1 being extremely bad (ie, more anxiety).
Subject comfort | 20 minutes
  Measured using a survey question asking participants to rank their comfort over the last 20 minutes using a scale of 5 being extremely positive; 4 being somewhat positive; 3 being neutral; 2 being somewhat negative; 1 being extremely negative

CONTACTS AND LOCATIONS:
Overall Officials: Suraj Kapa, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials